CLINICAL TRIAL: NCT03874273
Title: Targeted Therapy in Children and Adolescents With Recurrent, Progressive and Unresectable Inflammatory Myofibroblastic Tumor With the Inhibitor of Tyrosine Kinase -Crizotinib
Brief Title: Study of Crizotinib in Children and Adolescents With Myofibroblastic Tumors
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCPHOI-2019-01
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Inflammatory Myofibroblastic Tumor
Keywords: inflammatory myofibroblastic tumor; crizotinib; Paediatric oncology
MeSH Terms: conditions — Granuloma, Plasma Cell | interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- crizotinib + (Experimental): Patients with unresectable, relapsed or refractory inflammatory myofibroblastic tumor, receiving crizotinib
  Interventions: Drug: Crizotinib

INTERVENTIONS:
Drug: Crizotinib — Crizotinib 280mg/m2 twice a day (for 24 months maximum)
  Other Names: Xalkori

SUMMARY:
Targeted therapy based on target identification by genetic examinations is a promising direction in the treatment of patients with a complicated course of inflammatory myofibroblastic tumor. Recently, the main work covered in foreign publications, aimed at finding additional methods of treatment, by identifying new targets for targeted therapy in patients with unresectable IMT, but currently there is no standardized approach to the treatment of IMT in children worldwide.

This study can show the benefits of the usage of crizotinib as targeted therapy in children with ALK/ROS1 positive unresectable, progressive or reccurent inflammatory myofibroblastic tumors. The main hypothesis is that crizotinib would increase an objective response rate in this group of patients.

DETAILED DESCRIPTION:
Inflammatory myofibroblastic tumor (IMT) is a rare type of childhood neoplasm characterized by intermediate biological behavior. The main method of treatment of this tumor is a complete surgical removal. It should be said, that in 2-5% of patients the presence of distant metastases was noted at the time of diagnosis, in addition, the complex anatomical localization of the process sometimes does not allow a radical surgical intervention. In patients with unresectable IMT, the presence of distant metastases, residual tumor after initial resection or progression of the disease, attempts have been made to prescribe therapy with steroids , nonsteroidal anti-inflammatory drugs (NSAIDs), cytostatic drugs. However, the effectiveness of this therapy was low.

Since the late 90s, it is known that with the identification of a number of specific cytogenetic changes, this type of neoplasm is a true neoplastic process. In 50% of all cases of IMT there are clonal translocations of the ALK gene located at the 2p23 encoding the anaplastic lymphoma kinase (ALK). It was shown that ALK gene activation is based on translocations involving a large number of partner genes with tyrosine kinase activity. Currently, there are more than 21 partner genes involved in the formation of chimeric transcripts. The most frequent are TPM3, TPM4, CLTC, CARS, RANBP, EML4, TFG.

The introduction of modern molecular genetic methods, including the next generation sequencing (NGS), has expanded the understanding of the mechanisms of carcinogenesis in IMT. Along with ALK gene rearrangements, the ROS1 gene (YWHAE-ROS1 and TFG-ROS1) and PDGFRB (NAB2) genes were detected in the group of patients with ALK-negative IMT.

The therapy with tyrosine kinase inhibitors (crizotinib) has become possible not only in patients with ALK-positive tumor, but also in a group of patients who do not have an ALK gene rearrangement, but in whom a rearrangement of the ROS1 gene has been detected [4].

Previously, large-scale studies using tyrosine kinase inhibitors (crizotinib) have not been conducted in patients under 18 with IMT.

The Phase 1 study, conducted by the Children's Cancer Group (USA), showed the response rate on therapy with crizotinib in 3/7 patients, and . disease stabilization in 4/7 patients (Mosse Y., 2013).

The median age of patients with IMT, included in the study, was 8.4 years (range 1.1 - 21.4). In this study, it was noted that the use of crizotinib in a dose regimen of 280 mg / m2 twice a day in this group of patients does not lead to an increase in the incidence of side effects of grade 3 and 4. Thereby, the maximum permissible dose was determined, which amounted to 560 mg / m2 / day in two doses.

In the phase 2 study, it was shown that in the group of patients with IMO a response in 86% of cases has been achieved, with complete response in 36% (5/14), partial response in 50% (7/14), and stabilization of the disease in 14% (Mosse Y., 2017).

In the recently published single-drug, open-label, non-randomized phase 2 study the objective response rate on crizotinib in ALK+ patients was 50% (n=6/12) Schöffski P., et al. Lancet Respir Med. 2018 Jun;6(6):431-441. doi: 10.1016/S2213-2600(18)30116-4. Epub 2018 Apr 15).

The investigator's study is designed in order to show if the treatment with ALK-inhibitor crizotinib is able to improve the outcome of pediatric IMTs in Russia.

ELIGIBILITY:
Inclusion Criteria:

* Age 0 - 18 years
* The presence of a histologically verified diagnosis of Inflammatoru Myofibroblastic Tumor, confirmed in the pathology laboratory of Dmitry Rogachev National Research Center
* The presence of ttumor masses according to CT or MRI at the time of inclusion in the protocol
* Unresectable or metastatic tumor
* Relapse or progressive disease
* Good perfomance status
* Normal function of bone marrow
* Normal function of a liver
* Normal levels of creatinine and urea in blood
* Nornal heart funсtion (LVEF > 60%)
* Clear expression of rearranged ALK/ROS1 genes
* Signed Informed Consent

Exclusion Criteria:

* Age >18 years
* Refusal of signing the form of the informed consent
* The presence of comorbidities, which may endanger patient safety
* No rearrangements of ALK/ROS genes
* No signs of existing tumor, according to CT and MRI

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 2 months
  The frequency of response to therapy with Crizotinib in patients with translocation of the ALK / ROS1 genes and their partners.

SECONDARY OUTCOMES:
Relapse-free survival | 5 years
  Time after treatment without any signs or symptoms of inflammatory myofibroblastic tumor
Overall survival | 5 years
  The length of time from the start of treatment with crizotinib, that patients diagnosed with the inflammatory myofibroblastic tumor are still alive

CONTACTS AND LOCATIONS:
Locations (1):
- Dmitry Rogachev National Research Center of Pediatric Hematology, Oncology and Immunology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No